CLINICAL TRIAL: NCT03881449
Title: A Multicenter, 52-week, Provider- Randomized, Pragmatic Trial to Assess the Differences in ABILIFY MYCITE - a Digital Medicine System (DMS) Versus Treatment as Usual (TAU) for Adults With Schizophrenia, Bipolar I Disorder, or Major Depression Currently Using Aripiprazole
Brief Title: DIMES - DIgital MEdicine Study for Adults With Schizophrenia, Bipolar I Disorder, or Major Depression Currently Using Aripiprazole
Acronym: DIMES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Collaborators: Otsuka Pharmaceutical Development and Commercialization, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02188
Record Dates: First submitted 2019-02-19; First posted 2019-03-19 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Schizophrenia; Major Depressive Disorder; Bi-Polar Disorder; Schizo Affective Disorder
Keywords: digital medicine
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is an open-label 2-site (Durham and Houston Veterans Affairs (VA) Health Care Systems), provider randomized, prospective 2-arm (intervention vs. TAU) pragmatic trial. We will enroll 300 adult patients with schizophrenia, bipolar I disorder, or major depressive disorder currently being treated with oral Aripiprazole from either the Durham, North Carolina or Houston, Texas Veterans Affairs (VA) Health Care System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ABILIFY MYCITE Group (Experimental): If patients are assigned to the ABILIFY MYCITE treatment group, the patients and physician will initiate the system at the baseline visit, and continue to use the system for 3 months. At any time after the first 3 months, a patient and his or her doctor will have the opportunity to either discontinue or continue using ABILIFY MYCITE for the remainder of the trial (9 additional months; 12 months total) as long as clinically appropriate with the goal of measuring adherence to improve clinical decision-making and care.
  Both ABILIFY MYCITE and TAU participants will complete a battery of questions related to quality of life, patient usability/satisfaction, etc. at baseline, 3, 6 and 12 months.
  Interventions: Combination Product: ABILIFY MYCITE
- Treatment as Usual (TAU) Group (No Intervention): TAU patients will continue receiving care as recommended by their physician which will include the use of Aripiprazole according to the approved labels.
  Both ABILIFY MYCITE and TAU participants will complete a battery of questions related to quality of life, patient usability/satisfaction, etc. at baseline, 3, 6 and 12 months.

INTERVENTIONS:
Combination Product: ABILIFY MYCITE — Initiation of ABILIFY MYCITE will commence immediately, with subjects wearing the patch and using the smartphone app for a total of 3 months from baseline visit to the 3 month visit. Following the initial 90-days, the physician and patient may determine to use ABILIFY MYCITE anytime during the following 9 months. Following this period (up to 12 months), the subjects will not use ABILIFY MYCITE and return to standard care. A safety follow-up phone call will occur at 2 weeks after the 12 month/early termination (ET) visit. In addition, individuals in the ABILIFY MYCITE arm will evaluate satisfaction with the use of ABILIFY MYCITE.
  Arms: ABILIFY MYCITE Group

SUMMARY:
This is a 12 month, pragmatic trial designed to assess the differences in a digital medicine system (DMS)- ABILIFY MYCITE (Aripiprazole tablets with sensor)- measuring adherence versus treatment as usual (TAU) for adult patients with schizophrenia, bipolar I disorder, and major depression. Outcomes of interest will be adherence as measured by refill rates and all-cause and psychiatric health care use. Each patient will be in the study for a duration of 12 months.

All treatment medication decisions will be made by the healthcare professionals (HCPs) and not by protocol. Psychiatrist(s), nurse(s) and/or team manager(s) who will be responsible for subjects' care, will be considered as HCPs in this trial.

DETAILED DESCRIPTION:
This is a phase 4, 12-month, pragmatic trial designed to assess adherence in patients using ABILIFY MYCITE versus patients receiving treatment as usual (TAU). Both groups will complete surveys at baseline, 90, 180, and 360 days and will receive care at the discretion of their physician. The usual care group will not receive the ABILIFY MYCITE intervention. The primary outcome will assess refill rates at 6 months.

Eligible patients will enroll at their screening/baseline visit and ABILIFY MYCITE onboarding will be provided in the clinic, with commercial informational materials and additional call center support. Patients will then initiate 3 months of treatment with ABILIFY MYCITE at the baseline visit. At the Day 90 visit, patients will have the opportunity to either stop or continue using ABILIFY MYCITE for the remainder of the study (9 months). This decision must be a joint decision with the patient and his or her treating physician. During this optional interventional phase, patients may start and stop ABILIFY MYCITE as clinically indicated.

All enrolled patients will have required in-person visits at baseline, 90-days, and 180-days. The day 360 (final) visit can be in-person or via telephone.

Medical and actual pharmacy dispensing data will be collected from day 1 through day 360 using the VA's electronic medical record system.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years of age or older.
* Patients with a primary diagnosis of schizophrenia (including schizoaffective disorder), bipolar I disorder, or major depressive disorder based on the Diagnostic Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria.
* Patients have an active prescription for oral Aripiprazole.
* Patients may have general medical conditions that are deemed safe for the patient to enter an interventional trial per investigator judgment.
* Patients deemed fit for participation in the study by verbal or written confirmation from their mental health provider

Exclusion Criteria:

* Patients with a current neurocognitive disorder (i.e. dementia), intellectual disorder, or any other diagnosis that could impact the patient's ability to participate in the trial.
* Any patient who, in the opinion of the patient's mental health provider, study physician or investigator, is unfit to participate in the trial.
* Any patient who has participated in an investigational drug trial 30 days prior to trial enrollment.
* Females who are breastfeeding, and/or who have a positive pregnancy test prior to trial enrollment, or females who are planning to become pregnant during the trial. No clinical trials have been conducted on the use of ABILIFY MYCITE during pregnancy or breastfeeding.
* Patients who do not have skin on the anterior chest just above the lower edge of the rib cage that is free of any dermatological problems (e.g., dermatosis or dermatitis, open wounds, or other skin disorders such as warts, rashes, atopic dermatitis, or irritations).
* Patients who are unwilling to refrain from the use of topical products on the skin patch sites.
* Has 2 or more errors on the brief, 6-item cognitive screener administered at baseline.
* <20% Proportion of Days Covered (PDC) Aripiprazole over the last 6 months prior to enrollment. This is to ensure that all individuals enrolled will have at least filled their Aripiprazole prescription.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Aripiprazole refills | 6 months
  Aripiprazole refill as operationalized as a continuous measure of the number of days covered over the baseline to 6 month period

SECONDARY OUTCOMES:
Population Proportion of Days Covered (PDC) | 12 months
  The secondary outcomes of medication adherence (to Aripiprazole and other psychotic medications), defined as a binary indicators that PDC ≥ 80% for the prior 30-day period, are collected at baseline, 3, 6, and 12 months.
Days in acute care settings | 12 months
  The measure of days in acute care (i.e., days not in the community) over the 12-month outcomes interval defined as the total number of days in the ED or inpatient ward.

CONTACTS AND LOCATIONS:
Overall Officials: Hayden Bosworth, PhD, Principal Investigator — Durham VA Medical Center
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, North Carolina
  - Michael E. DeBakey VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzales S, Okusaga OO, Reuteman-Fowler JC, Oakes MM, Brown JN, Moore S, Lewinski AA, Rodriguez C, Moncayo N, Smith VA, Malone S, List J, Cho RY, Jeffreys AS, Bosworth HB. Digital Medicine System in Veterans With Severe Mental Illness: Feasibility and Acceptability Study. JMIR Form Res. 2022 Dec 22;6(12):e34893. doi: 10.2196/34893. PMID 36548028